CLINICAL TRIAL: NCT06173635
Title: A Laboratory Trial to Explore the Benefits of the New Maxi Move 5 (MM5) Technology
Brief Title: A Comparison Study of the Maxi Move 5 (MM5) Device
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Arjo AB (Industry)
Collaborators: Loughborough University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: MaxiMove5-MACC-001-2023
Record Dates: First submitted 2023-10-23; First posted 2023-12-18 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-08

CONDITIONS: Healthy Volunteers

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Maxi Move 5 (Other): 24 healthy volunteers will evaluate all 5 devices
  Interventions: Device: Maxi Move 5

INTERVENTIONS:
Device: Maxi Move 5 — 4 comparative devices will be used to evaluate the MM5 device

SUMMARY:
This trial aims to evaluate the added improvements from a caregiver and patient benefit perspective.

The trial should identify the forces involved for the caregiver when manoeuvring the lift.

ELIGIBILITY:
Inclusion Criteria:

For expert patient:

* ≥18 years
* Healthy male or female
* 80-100 kg

  24 healthy volunteers (caregivers) will be recruited. They will require a strong working knowledge of passive floor lifts and patient positioning with the use of loop and clip slings.

Exclusion Criteria:

-

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2023-12-20 (Actual); Primary Completion 2024-02-28 (Actual); Study Completion 2024-05-31 (Actual)

PRIMARY OUTCOMES:
1. Time to complete each transfer will be recorded | up to 24 months
  Time to complete each activity and each task within the activity will be measured in seconds.
2. A detailed hierarchical task analysis (HTA) of each activity will be completed using the video recordings and experimenter field notes for each transfer to asses the number of correct placements for each device. | up to 24 months
  Correct placement will be visually controlled with the use of markers on the subject and the final positioning device (e.g chair, toilet or bed) for each transfer. This will be reported as distance from the ideal position.
3. Physical load for movement of the hoist throughout the activities for each device will be measured. | up to 24 months
  Force required to complete the range of patient and hoist positioning tasks, forward, backwards, rotation movement, patient positioning etc. These forces will be used with the HTA data to calculate the amount of physical force delivered by the participants with each device and each transfer. The forces used will be presented in newton.
4 Collect subjective data from the caregivers that describe, comfort, ease of use, effort and willingness to adopt in practice, etc | up to 24 months
  This will be collected by the use of questionnaires
5 Subjective responses from the expert patient being transferred will be recorded | up to 24 months
  This will be collected by the use of questionnaires

CONTACTS AND LOCATIONS:
Overall Officials: Karin Hannander, Study Director — Arjo AB
Locations (1):
- School of Design and Creative Art at Loughborough University, Loughborough, United Kingdom